CLINICAL TRIAL: NCT01317940
Title: Nutrition and Body Composition in Acute Lymphoblastic Leukemia (Environment and Microenvironment in ALL #2)
Brief Title: Nutrition and Body Composition in Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Etan Orgel, Clinical Fellow, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCI-10-00273; LLS 6249-11 (Other Grant/Funding Number: Leukemia and Lymphoma Society)
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma; Vitamin D Deficiency
Keywords: Leukemia; ALL; Vitamin D; Bone Density; Body Fat; Obesity; Adipose
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Vitamin D Deficiency; Leukemia; Obesity | interventions — Vitamin D; Calcium Citrate; Calcitriol; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Newly Diagnosed Subjects) (Experimental)
  Interventions: Dietary Supplement: Vitamin D and Calcium Citrate
- Standard of Care Group A (No Intervention)
- Group B (Early Survivors) (Experimental)
  Interventions: Dietary Supplement: Vitamin D and Calcium Citrate
- Observation Only - Group B (No Intervention)
- Group C (Siblings of Group A) (No Intervention)

INTERVENTIONS:
Dietary Supplement: Vitamin D and Calcium Citrate — Vitamin D (10,000 int.units/ml) 100,000 int. units (10ml) by mouth once every two months x 3 times (total treatment period approximately 6-7 months)
  Calcium Carbonate (1,000 mg/tab = 400 mg elemental calcium/tab) 2,000 mg (2 chewable tabs) by mouth every day for approximately 6-7 months
  Other Names: 1,25-Dihydroxycholecalciferol; Calcitriol; Rocaltrol (Roche); Calcium carbonate
  Arms: Group A (Newly Diagnosed Subjects); Group B (Early Survivors)

SUMMARY:
Many adolescents with acute lymphoblastic leukemia (ALL) have been found to have low bone density by the end of treatment. This can lead to long-term suffering in survivors due to poor bone health. Vitamin D is known to be associated with bone health and previous research has established that Vitamin D insufficiency is very common at diagnosis of ALL and worsens over the course of treatment. Researchers have also learned that a relationship exists between both Vitamin D and fat tissue and ALL and fat tissue.

In adolescents being treated for ALL as well as in early survivors, this randomized study will therefore examine the effect of Vitamin D and calcium supplementation on correcting Vitamin D insufficiency and on improving bone density in the context of changes in body composition and body fat. Bone density will be measured by a radiology exam called qCT (quantitative computed tomography) while body composition and body fat will be measured by a different radiology exam called a DXA (dual energy x-ray absorptiometry scan) . The study will also examine in depth the relationship between these three elements - Vitamin D insufficiency, obesity, and ALL - and their impact on bone density.

ELIGIBILITY:
Inclusion Criteria:

GROUP A: Patients with newly diagnosed ALL

* Are greater than or equal to 10 years of age and less than or equal to 21 years of age at diagnosis of ALL
* Have a new diagnosis of untreated ALL classified as "high risk" per NCI criteria (due to being greater than 10 years of age)
* Are beginning treatment with a Children's Cancer Group/Children's Oncology Group "high risk" protocol with a 4-drug induction including steroids
* Are not pregnant

GROUP B: Early survivors of ALL

* Were treated for ALL and remain in first CR1 (complete remission)
* Were equal to or greater than 10 years of age and less than or equal to 21 years of age at diagnosis of ALL
* Have completed treatment on or as per a Children's Cancer Group/Children's Oncology Group "high risk" protocol between 12 and 48 months prior to enrollment in this study (consisting of a plan for a 4-drug induction including steroids in Induction, Delayed Intensification, and steroid pulses in Maintenance. Steroids are allowed to have been discontinued due to toxicity).
* Are not pregnant

GROUP C: Siblings of Group A

* Are either a full-sibling or a half-sibling of a patient in Group A
* Are living at the same residence as the sibling/half-sibling from Group A
* Are greater than or equal to 10 years of age and less than or equal to 21 years of age at the time of study entry, and within 3 years of the age diagnosis of ALL in the sibling/half-sibling from Group A
* Are on the same Vitamin D supplementation regimen (if any) as the sibling from Group A at the time of his or her diagnosis

Exclusion Criteria (All Groups):

* Have a diagnosis of Down syndrome (Trisomy 21) or any genetic disease associated with abnormal bone development
* Are undergoing treatment with other medicines that affect bones including chronic use of of steroids, bisphosphonate therapy, or Vitamin D at average dose greater than 400 international units (IU)/day
* Have an underlying diseases altering body structure (i.e. missing a limb, severe dysmorphism) or severely affecting mobility (i.e. total or hemiparesis)
* Have a history of chemotherapy or radiation for other cancers
* Cannot complete the radiology exams/radiology exams uninterpretable (i.e. people with a hip replacement or prosthesis)

Ages: 10 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Etan Orgel, MD, Principal Investigator — Children's Hospital Los Angeles; Steven Mittelman, MD, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Orgel E, Framson C, Buxton R, Kim J, Li G, Tucci J, Freyer DR, Sun W, Oberley MJ, Dieli-Conwright C, Mittelman SD. Caloric and nutrient restriction to augment chemotherapy efficacy for acute lymphoblastic leukemia: the IDEAL trial. Blood Adv. 2021 Apr 13;5(7):1853-1861. doi: 10.1182/bloodadvances.2020004018. PMID 33792627
- See also: NIH Vitamin D Fact Sheet — http://ods.od.nih.gov/factsheets/vitamind/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Group A: 2 participants enrolled but did not reach time of randomization (1 induction death, 1 severe toxicity/change in treatment plan) Group B: 2 subjects enrolled but did not reach time of randomization or undergo any study procedures (2 lost to follow-up)
Groups:
- On-Therapy Intervention (Group A): Subjects randomized following Induction to receive education plus:
  Vitamin D and Calcium Citrate: Vitamin D (10,000 int.units/ml) 100,000 int. units (10ml) by mouth once every two months x 3 times (total treatment period approximately 6-7 months) Calcium Carbonate (1,000 mg/tab = 400 mg elemental calcium/tab) 2,000 mg (2 chewable tabs) by mouth every day through study period (total treatment period approximately 6-7 months)P
- On Therapy Standard of Care (Group A): Subjects randomized following Induction to receive standard of care with education alone OR subjects ineligible for open-label randomization and followed as "natural history" cohort.
- On-Therapy "Natural History" (Group A): Patients enrolled prior to open-label randomization and those not eligible for randomization at end of induction
- Survivorship Intervention (Group B): Subjects randomized to receive education plus directly-observed therapy with open-label Vitamin D and chewable calcium
- Survivorship Standard of Care (Group B): Survivors randomized to receive standard of care with education alone OR subjects ineligible for open-label Vitamin D+ Calcium randomization and continued with follow-up only.
- Siblings of Survivors (Group C): Healthy siblings of survivors of pediatric acute lymphoblastic leukemia (ALL) for one-time assessment
Period: Overall Study
Arm/Group | On-Therapy Intervention (Group A) | On Therapy Standard of Care (Group A) | On-Therapy "Natural History" (Group A) | Survivorship Intervention (Group B) | Survivorship Standard of Care (Group B) | Siblings of Survivors (Group C)
Started | 19 | 10 | 20 | 6 | 13 | 4
Completed | 18 | 10 | 15 | 5 | 12 | 4
Not Completed | 1 | 0 | 5 | 1 | 1 | 0
Not completed — Death | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Change in therapy plan | 0 | 0 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- On Therapy Intervention (Group A): Subjects randomized following Induction to receive education plus:
  Vitamin D and Calcium Citrate: Vitamin D (10,000 int.units/ml) 100,000 int. units (10ml) by mouth once every two months x 3 times (total treatment period approximately 6-7 months) Calcium Carbonate (1,000 mg/tab = 400 mg elemental calcium/tab) 2,000 mg (2 chewable tabs) by mouth every day through study period (total treatment period approximately 6-7 months)P
- On Therapy Standard of Care (Group A): Subjects randomized following Induction to receive standard of care with education alone
- On Therapy "Natural History" (Group A): Subjects surviving to end of Induction but ineligible for randomization for any reason
- Survivorship Intervention (Group B): Survivors to receive education plus:
  Vitamin D and Calcium Citrate: Vitamin D (10,000 int.units/ml) 100,000 int. units (10ml) by mouth once every two months x 3 times (total treatment period approximately 6 months) Calcium Carbonate (1,000 mg/tab = 400 mg elemental calcium/tab) 2,000 mg (2 chewable tabs) by mouth every day through study period (total treatment period approximately 6 months)
- Survivorship Standard of Care (Group B): Survivors either randomized to received standard of care with education alone OR vitamin D sufficient and continued for follow-up only.
- Siblings (Group C): Healthy siblings of subjects in Group A
- Total: Total of all reporting groups
Arm/Group | On Therapy Intervention (Group A) | On Therapy Standard of Care (Group A) | On Therapy "Natural History" (Group A) | Survivorship Intervention (Group B) | Survivorship Standard of Care (Group B) | Siblings (Group C) | Total
Number analyzed (Participants) | 19 | 10 | 20 | 6 | 13 | 4 | 72
Age, Continuous [Median (Full Range); unit: years] | 15 [11 to 19] | 15 [11 to 18] | 14 [10 to 19] | 19 [16 to 21] | 18 [15 to 23] | 15 [12 to 21] | 15 [10 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 9 | 3 | 3 | 4 | 29
  Male | 13 | 6 | 11 | 3 | 10 | 0 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 8 | 16 | 5 | 5 | 3 | 54
  Not Hispanic or Latino | 2 | 2 | 4 | 1 | 3 | 0 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 19 | 10 | 20 | 6 | 13 | 4 | 72

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Vitamin D Level (Group A)
Description: Change in Vitamin D levels from baseline to study end (Group A: Consolidation through end of Delayed Intensification)
Time Frame: +6 months
Population: Includes subjects in each group evaluable for vitamin D endpoint. Calculation of change = Vitamin D level at study end (end of DI, ~+6 months)/Vitamin D level at baseline (start of consolidation).
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | On-Therapy Intervention (Group A) | On Therapy Standard of Care (Group A) | On-Therapy "Natural History" (Group A)
Number analyzed (Participants) | 18 | 10 | 15
ng/ml
  Change in serum Vitamin 25(OH)D level | 5.5 (1.7) | -0.30 (2.2) | 1.0 (2.6)
  Post-intervention serum Vitamin 25(OH)D level | 26.5 (12.4) | 19.0 (7.4) | 23.3 (2.8)

2. Secondary Outcome: Bone Mineral Density by Quantitative Computed Tomography (QCT) at Study End (Group A)
Description: Bone mineral density (vBMD) at end of study period (Group A: end of Delayed Intensification)
Time Frame: +6 months
Population: Subjects enrolled following the change to the open-label randomization were imaged for cortical bone density at the femur, subjects enrolled prior to this in the Natural History group were imaged at the tibia. The change was made for later subjects due to technical reasons to provide a better estimate of cortical density.
Measure: Mean (Standard Deviation); unit: cm3
Groups:
- On-Therapy "Natural History" (Group A, Tibia): Patients enrolled prior to open-label randomization and those not eligible for randomization at end of induction
Arm/Group | On-Therapy Intervention (Group A) | On Therapy Standard of Care (Group A) | On-Therapy "Natural History" (Group A, Tibia)
Number analyzed (Participants) | 17 | 10 | 14
cm3
  Cortical BMD | 2093.1 (62.5) | 2090.9 (26.7) | 927.5 (65.3)
  Cancellous BMD | 203.8 (77.1) | 201.4 (66.4) | 159.1 (54.9)

3. Secondary Outcome: Change in Vitamin D Level (Group B)
Description: Change in serum vitamin D level was assessed in survivors at baseline and after 6 months of supplementation
Time Frame: +6 months
Population: Change in Vitamin D = Vitamin D at +6months/Vitamin D at baseline
Measure: Median (Standard Error); unit: ng/ml
Arm/Group | Survivorship Intervention (Group B) | Survivorship Standard of Care (Group B)
Number analyzed (Participants) | 5 | 12
ng/ml
  Change in serum Vitamin 25(OH)D level | 1.0 (2.2) | -1.0 (2.1)
  Post-intervention serum Vitamin 25(OH)D level | 26.0 (2.0) | 29.0 (2.9)

4. Secondary Outcome: Bone Mineral Density by QCT in Survivors at Study End (Group B)
Description: Bone mineral density (vBMD) at end of study period (Group B: after 6 months)
Time Frame: +6 months
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | Survivorship Intervention (Group B) | Survivorship Standard of Care (Group B)
Number analyzed (Participants) | 5 | 7
cm3
  Cortical bone mineral density | 2087.4 (39.3) | 2049.3 (73.0)
  Cancellous bone mineral density | 243.6 (28.7) | 269.3 (80.0)

5. Secondary Outcome: Prevalence of Obesity and Vitamin D Insufficiency in Adolescents With Newly Diagnosed ALL and in Their Siblings
Description: Insufficiency defined as 25(OH)D < 30 ng/ml
Time Frame: 1 timepoint
Population: Group C: Only four siblings enrolled and arm closed early due to poor accrual. Specimens from this group were not analyzed so no results are available.
  Group A: 39 subjects enrolled at diagnosis had Vitamin D testing performed at diagnosis and had results available.
Measure: Count of Participants; unit: Participants
Groups:
- Siblings of Survivors (Group C): Healthy siblings of survivors of pediatric ALL for one-time assessment
- Newly Diagnosed Patients (Group A): Siblings enrolled in trial (Group A)
Arm/Group | Siblings of Survivors (Group C) | Newly Diagnosed Patients (Group A)
Number analyzed (Participants) | 0 | 39
Participants | 0 | 36

ADVERSE EVENTS:
Time Frame: 6 months (Randomization to end of study)
Description: Note that subjects in the On-Therapy "natural history" arm (i.e. Group A, not randomized) were not formally followed for adverse event reporting.
  Subjects in Sibling group (Arm C) had a single visit for a laboratory draw with no adverse event reporting indicated.
Groups:
- On Therapy Intervention (Group A): Subjects randomized following Induction to receive education plus:
  Vitamin D and Calcium Citrate: Vitamin D (10,000 int.units/ml) 100,000 int. units (10ml) by mouth once every two months x 3 times (total treatment period approximately 6 months) Calcium Carbonate (1,000 mg/tab = 400 mg elemental calcium/tab) 2,000 mg (2 chewable tabs) by mouth every day through study period (total treatment period approximately 6 months)
- Survivorship Intervention (Group B): Survivors randomized to receive directly-observed therapy with open-label Vitamin and chewable calcium
- Survivorship Standard of Care (Group B): Survivors randomized to receive standard of care with education alone OR ineligible for open-label Vitamin D+Calcium randomization
- Siblings of Group A (Group C): Singling of Group A were enrolled for a one-time visit for labs; All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | On Therapy Intervention (Group A) | On Therapy Standard of Care (Group A) | Survivorship Intervention (Group B) | Survivorship Standard of Care (Group B) | Siblings of Group A (Group C)
All-Cause Mortality (participants affected / at risk) | 1/19 | 0/10 | 0/6 | 0/13 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/10 | 0/6 | 0/13 | 0/0
Other Adverse Events (participants affected / at risk) | 0/19 | 0/10 | 0/6 | 0/13 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No